CLINICAL TRIAL: NCT06622551
Title: The Study of Association Between Obesity and Iron Deficiency Anaemia in Nonpregnant Indonesian Women
Brief Title: Different Efficacy of IFA Supplementation Among Obese and Non-obese Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Griffith University (Other)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Qonita Rachmah, Principle Investigator, Griffith University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GU Ref No: 2024/228; 3433/BPPT/BPI.LG/V/2024 (Other Grant/Funding Number: BPI Kemdikbud); 119/EA/KEPK/2024 (Other: KEPK FKM UNAIR); U1111-1313-7880 (Other: Universal Trial Number)
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Overweight; Anemia, Iron-Deficiency
Keywords: Obesity; Iron folic acid supplemet; Anemia; Women of reproductive age; Indonesia
MeSH Terms: conditions — Obesity; Overweight; Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Overweight/obese arm (Experimental): In this arm, those who are overweight and obese will be assigned. Each participant will be given 90 days of IFA supplement.
  Interventions: Dietary Supplement: Iron-folic acid supplement
- Normal-weight arm (Active Comparator): In this arm, those with normal-weight will be assigned. Each participant will be given 90 days of IFA supplement.
  Interventions: Dietary Supplement: Iron-folic acid supplement

INTERVENTIONS:
Dietary Supplement: Iron-folic acid supplement — The major thing distinguishing this clinical study from another clinical trial is that we differentiate intervention based on nutritional status as we want to observe whether different nutritional status, especially overweight/obese will diminish the effect of IFA supplementation.

SUMMARY:
This clinical trial aims to learn if there is a relationship between OWT/OB and IDA in nonpregnant women of reproductive age and its impact on iron supplementation. The main questions it aims to answer are:

* Is there any independent association between overweight/obesity and iron deficiency anemia in nonpregnant women after controlling for potential confounding factors?
* Does the effect of iron supplementation on iron status vary between overweight/obese and normal-weight nonpregnant women (as measured by multiple iron biomarkers)? Researchers will compare several biomarkers between the case and control groups after the intervention is given for 90 days.

Participants will:

* Visit the research center before the intervention given and after 90 days
* Take daily iron-folic acid supplements for 90 days
* Keep a diary of their supplement's intake

DETAILED DESCRIPTION:
Anaemia is one of the major nutritional problems that brings many negative health consequences to women's health, especially during pregnancy. There was growing evidence that overweight/obesity can lead to anaemia. However, the association between anaemia and overweight/obesity has not been fully established, especially in developing countries, including Indonesia. The prevalence of overweight/obesity has sharply increased in Indonesia for the past decades, while anaemia prevalence did not show a significant decrease. The prevalence of anaemia in Indonesia was still alarming, with 27.2% in nonpregnant women and 48.9% in pregnant women (Indonesia MoH, 2019a). Therefore, the study of the association between overweight/obesity and anaemia among women of reproductive age in Indonesia needs to be conducted using appropriate measurements. Furthermore, previously available studies highly ignored the role of dietary intake in the association between overweight/obesity and anaemia despite its importance. This study will also measure dietary intake among women.

Once participants agree to participate in this study, the investigators will ask questions about themselves (latest education history, employment, general health, menstrual history, smoking history, and physical activity level). The investigators will then ask the participants to write the food and beverages consumed in the dietary record form for 3-non consecutive days. Then, the investigators will ask about their dietary intake in the last 24 hours/1 day (foods the participants have taken and their approximate amount). After that, the investigators will take anthropometric measurements (height, weight, and waist circumference) to define nutritional status. The investigators will also collect a small amount (3mL) of blood samples from the participants, two times (before and after intervention). Blood collection will be performed by trained nurses/medical analysts under a medical doctor's supervision and collected at the university clinic. The investigators will measure several parameters from that blood sample, such as iron status parameters (including hemoglobin, serum ferritin, and hepcidin) and other chemicals in the blood that indicate inflammation (AGP and CRP). The results of these tests will be provided to all participants.

After collecting these data, participants will be assigned to one of the two study groups using matching criteria (age, education level, and occupation). Participants in all groups will receive iron supplements. The participants will not be made aware of which arm they have been assigned to. For the following three months, the participants will receive approximately 90 iron supplements to be consumed every day. The study staff will contact the participants through short messages and monthly visitation to ensure adherence to iron supplement consumption. After three months, the investigators will stop providing iron supplements. The investigators will collect information about their dietary intake over the last day and retake their anthropometry measurements. The investigators will also collect blood samples from participants and perform the same test as the previous one.

The investigators have asked the subjects to participate in this study because the participants are women aged between 20 and 29 years, neither pregnant nor lactating, living in this area, are healthy, have not received any micronutrient supplementation in the last three months, and have not undergoing body mass reduction or on any particular weight loss diet. After anthropometric screening, each participant will be assigned to a case or control group based on the Body Mass Index (BMI) results.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant, nonlactating women aged 19 - 29 years
* Never been married and pregnant.
* Having no menstrual abnormality (amenorrhea, polymenorrhea, etc.)
* Able to read and write in Bahasa Indonesia
* Not undergoing body mass reduction or on any particular weight loss diet

Exclusion Criteria:

* BMI <18.5 kg/m2
* Self-reported specific diseases that need diet modification (i.e., type 1 diabetes, kidney disease, autoimmune disease, etc.)
* Self-report of significant medical conditions (e.g., diabetes mellitus, disorders of the liver [including hemochromatosis] and kidney, autoimmune or metabolic diseases, and malignancy] or use of medications that may influence weight, iron, or inflammatory status; pregnancy or lactation; vegetarianism; zinc supplementation; smoking habit.

Ages: 20 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Iron Deficiency Anemia (IDA) | From enrollment to the end of treatment at 90 days
Concentration of Hemoglobin | Day 0 (Before intervention) and Day 90 (After intervention)
  Concentration of Hb will be measured in g/dL
Concentration of Ferritin | Day 0 (Before intervention) and Day 90 (After intervention)
  Aims to assess iron deficiency among women; will be measured in ng/mL
Concentration of Hepcidin | Day 0 (Before intervention) and Day 90 (After intervention)
  Concentration of Hepcidin will be measured in ng/mL
Overweight and obese prevalence | Day 0 (Before intervention) and Day 90 (After intervention)
  To achieve this outcome, weight will be measured in Kilograms and height will be measured in centimeters. Weight and height will be combined to report BMI in kg/m^2.
Concentration of CRP | Day 0 (Before intervention) and Day 90 (After intervention)
  The concentration of CRP will be measured in mg/L
Concentration of AGP-1 | Day 0 (Before intervention) and Day 90 (After intervention)
  The concentration of AGP-1 will be measured in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Ahmed, Convenor, Study Director — Griffith University
Locations (1):
- Nutrition Laboratory, Faculty of Public Health Universitas Airlangga, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication. All data collected from participants will only be used for research or academic purposes, i.e., publishing an article in a research journal, presenting the findings in a conference or seminar, or teaching in the classroom. Participant name and contact details will not be shown when presenting the study findings in an article or a seminar.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting information will be available from January 2025 until the next 5 years.
Access Criteria: Only the study investigators from Griffith University (QLD, Australia) will have access to your personal information.